CLINICAL TRIAL: NCT02195440
Title: An Open Label, Single Arm, Dose Escalation Phase 1 Trial of PRI-724 in Patients With HCV-induced Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Komagome Hospital (Other)
Collaborators: Prism Pharma Co., Ltd. (Industry); Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Kiminori Kimura, MD, MD, Komagome Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRI-724-1101; UMIN000014395 (Other: UMIN (University Hospital Medical Information) CTR)
Record Dates: First submitted 2014-07-08; First posted 2014-07-21 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C Virus-infected Cirrhosis
Keywords: Hepatitis C virus, cirrhosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRI-724 (Experimental): 3 cohorts (PRI-724: 10, 40, 160 mg/m2/day), 6 cycles (1 cycle: 1-week continuous i.v. administration+1-week observation period)
  *Cycle 2 will not be started until plasma drug concentrations of PRI-724 and C-82 on Days 1 and 2 in Cycle 1 are confirmed.
  Cohort 1: 10 mg/m2/day (6 subjects) Cohort 2: 40 mg/m2/day (6 subjects) Cohort 3: 160 mg/m2/day (6 subjects) One cycle consists of 1-week continuous i.v. administration of PRI-724 followed by a 1-week observation period. The tolerability and safety after 6 cycles will be confirmed.
  Interventions: Drug: PRI-724

INTERVENTIONS:
Drug: PRI-724 — 10 - 160 mg/m2, 7 days CIV (in the vein) with 7 days rest per one cycle. Number of Cycles: 6.
  Other Names: CBP-beta-catennin inhibitor; OP-724

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of PRI-724 in patients with HCV-induced cirrhosis.

DETAILED DESCRIPTION:
This is a single-center, open-label, continuous i.v. administration, dose escalation Phase I study in patients with hepatitis C cirrhosis.

One cycle consisted of one-week continuous i.v. administration of PRI-724 followed by a one-week observation period. One cohort was a total of six cycles, a 12-week treatment period.

PRI-724 was administered at a dose of 10 mg/m2/day in Cohort 1, 40 mg/m2/day in Cohort 2, and 160 mg/m2/day in Cohort 3 in a dose escalation manner. Each cohort was to include 6 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of cirrhosis due to hepatitis C virus. 1) Serum HCV-RNA test positive 2) Definitive diagnosis of cirrhosis established by liver biopsy (HAI score: Grade IV-D).
2. Child-Pugh Class A or B at the time of informed consent, with no likelihood of improvement with existing medical treatment.
3. Performance Status: 0 - 2.
4. Between =>20 and <75 years of age at the time of providing written consent.
5. Having provided voluntary written consent for participation in this study.
6. Esophageal and gastric varices are well controlled

Exclusion Criteria:

1. Patients with cirrhosis due to causes other than hepatitis C virus; or patients with cirrhosis due to unknown causes.
2. Patients with a history of primary liver cancer or a complication thereof.
3. Patients with a complication of malignant tumor or a history thereof (within 5 years prior to screening).
4. Patients in whom such active viral infections as HBV, HIV or ATCL or syphilis infection cannot be ruled out.
5. Patients with serum creatinine >1.5 times over upper normal or creatinine clearance =<60 mL/min/1.73 m2.
6. Patients with hemoglobin <8 g/dL.
7. Patients with platelet count <50,000 /&micro;L.
8. Patients with T.Bil =>3.0 mg/dL.
9. Patients with a complication of poorly controlled diabetes, hypertension or heart failure.
10. Patients with a complication of mental disorder requiring treatment.
11. Patients with serious allergy to contrast media or a history thereof.
12. Patients with allergy to inactive ingredients of the study drug.
13. Patients who have received interferon, ribavirin or anti-HCV agents within 12 weeks before registration in this study.
14. When the medical treatment to a primary disease is carried out, Patient who was changed the dosage and administration within the 12 weeks before registration.
15. Patients with a history of drug or alcohol addiction within five years at the time of providing written consent or a history of drug or alcohol abuse within the past one year.
16. The patient who received a liver transplant or other organ transplants (a bone marrow transplantation is included), and the patient for whom intravenous administration and venous access are difficult.
17. Patients contraindicated for liver biopsy.
18. Female patients who are pregnant or suspected to be pregnant; or those who desire to get pregnant during the study period or those of childbearing potential.
19. Male patients who do not consent to practice birth control during the clinical study.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events and adverse drug reactions (including subjective symptoms and abnormal laboratory values) | 12 weeks after the initiation of PRI-724 administration
  Items and ratio%

SECONDARY OUTCOMES:
Child-Pugh Score | 12 weeks after the initiation of PRI-724 administration
  Changes of score
Liver biopsy: Histology Activity Index (HAI) | 12 weeks after the initiation of PRI-724 administration
  Changes of index
Serum albumin level | 12 weeks after the initiation of PRI-724 administration
  Changes of level
Serum fibrosis marker level(s) | 12 weeks after the initiation of PRI-724 administration
  Changes of level
Ascitic fluid level | 12 weeks after the initiation of PRI-724 administration
  Changes of level
Improvement rate of lower leg edema | 12 weeks after the initiation of PRI-724 administration
  Changes of rate
Assessment of Area under the plasma concentration versus time curve (AUCinf) of PRI-724 through analysis of blood samples | Days 1-2 for preinfusion, 0.5, 1.0, 2.0, 4.0, and 24h; Day 7-8 for prestopping, 0.5, 1.0, 2.0, 4.0, and 24h
  Comparison of AUC
Assessment of Steady State Plasma Concentration (Css) of PRI-724 through analysis of blood samples | Days 1-2 for preinfusion, 0.5, 1.0, 2.0, 4.0, and 24h; Day 7-8 for prestopping, 0.5, 1.0, 2.0, 4.0, and 24h
  Comparison of Css

CONTACTS AND LOCATIONS:
Overall Officials: Kiminori Kimura, MD, Principal Investigator — Komagome Metropolitan Hospital
Locations (1):
- Tokyo metropolitan Komagome Hospital, Tokyo, Japan

REFERENCES:
- [Derived] Kimura K, Ikoma A, Shibakawa M, Shimoda S, Harada K, Saio M, Imamura J, Osawa Y, Kimura M, Nishikawa K, Okusaka T, Morita S, Inoue K, Kanto T, Todaka K, Nakanishi Y, Kohara M, Mizokami M. Safety, Tolerability, and Preliminary Efficacy of the Anti-Fibrotic Small Molecule PRI-724, a CBP/beta-Catenin Inhibitor, in Patients with Hepatitis C Virus-related Cirrhosis: A Single-Center, Open-Label, Dose Escalation Phase 1 Trial. EBioMedicine. 2017 Sep;23:79-87. doi: 10.1016/j.ebiom.2017.08.016. Epub 2017 Aug 19. PMID 28844410